CLINICAL TRIAL: NCT02341742
Title: Relationship Between Physical Activity and Bone Mineral Density in Children and Adolescents With Chronic Inflammatory Bowel Disease
Brief Title: Physical Activity and Bone Mineral Density in Children and Adolescents With Chronic Inflammatory Bowel Disease
Acronym: PHYSICOSMICI
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_69; 2014-A00685-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Physical activity; Bone health; Pediatrics; Bone
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: follow up of patients (children and adolescent) with inflammatory bowel disease in looking for the relationship between the bone mineral density and physical activity.
  Interventions: Device: multiple examinations

INTERVENTIONS:
Device: multiple examinations — biological,clinical, X-ray, DXA, accelerometry assessment

SUMMARY:
This study is an observational study. The purpose of this study is to assess the relationship between bone health and daily physical activity in children and adolescents with inflammatory bowel disease (IBD). Reduced bone mineral density is a common complication in pediatric IBD. Physical activity is an important determinant of health throughout the whole lifespan. Engaging in regular moderate-to-vigorous physical activity has important health benefits. Based on available evidence, the investigators hypothesize that daily moderate-to-vigorous physical activity could improve bone health (ie bone mineral density) in children and adolescents with IBD.

DETAILED DESCRIPTION:
To carry out this study, 120 patients (age ≥6 and <18 years at the screening visit) will be enrolled in this observational study. After obtaining the informed consent from the parents and the patient, the followings will be performed: clinical examination by a physician, dual-energy X-ray absorptiometry to assess bone density mineral and body composition, collection of a blood sample to assess the inflammatory status of the IBD patient. The patient will be asked also to fill in a questionnaire in order to assess quality of life. He will wear an accelerometer during 7 consecutive days for assessing daily physical activity in free living conditions. The main objective is to assess the relationship between daily physical activity and bone health in children and adolescents with IBD. The secondary objectives are to assess the relationship between daily physical activity and: 1) body composition and 2): quality of life in IBD children and adolescents. To our knowledge, this study is the first to assess the relationship between bone health and daily physical activity in IBD children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls aged between 6 and 18 years old
* Chronic, acute or intermittent diseas (other than IBD) that can lead to decreased physical activity (example: fracture, paralysis, blindness ...
* Patient with IBD diagnosed since at least 6 months
* Written informed consent obtained by the the parents and the patient
* To have a health insurance

Exclusion Criteria:

* Acute intercurrent events (less than 15 days) at the inclusion day leading to decreased physical activity according to the investigator judgment (fracture(s), recent arthritis, perineal lesions, severe skin lesions)
* Patient refusing to participate to the study
* One of the child's parents refusing to participate to the study
* Lack of adherence foreseeable
* Participation to another study
* Pregnant girls
* Under a justice protect measure

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and Adolescents With Inflammatory Bowel Disease: Crohn´s disease and Ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dual energy-ray absorptiometry (bone mineral density) | At 3 weeks
  We assess the bone mineral density with the Dual energy-ray absorptiometry method at the visit 2 corresponding at 3 weeks after the visit 1

SECONDARY OUTCOMES:
Dual energy-ray absorptiometry (Fat Mass) | At 3 weeks
  We assess the Fat Mass with the Dual energy-ray absorptiometry method at the visit 2 corresponding at 3 weeks after the visit 1
Dual energy-ray absorptiometry (Fat Free Mass) | At 3 weeks
  We assess the Fat Free Mass with the Dual energy-ray absorptiometry method at the visit 2 corresponding at 3 weeks after the visit 1
Accelerometry ( Physical Activity) | At 3 weeks
  We assess the Physical Activity with the accelerometry method during 7 consecutive days
IMPACT III Questionnaire (quality of life) | At 3 weeks
  We assess the quality of life throughout the IMPACT III questionnaire at the visit 2 corresponding at 3 weeks after the visit 1
PedsQL Questionnaire (quality of life) | At 3 weeks
  We assess the quality of life throughout the PedsQL questionnaire at the visit 2 corresponding at 3 weeks after the visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Dominique TURCK, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Clinical Investigation Center, Lille, Nord
  - Chu Amiens-Picardie - Site Sud, Amiens
  - Centre Hospitalier, Arras
  - Centre hospitalier, Béthune
  - Centre Hospitalier, Lens
  - Centre Hospitalier St Vincent, Lille
  - Centre Hospitalier, Roubaix

REFERENCES:
- [Derived] Vanhelst J, Beghin L, Drumez E, Djeddi-Dine D, Tuck D, Coopman S, Gottrand F, Ley D. Validation of the IMPACT-III Questionnaire in French Children With Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2023 Apr 1;76(4):e71-e76. doi: 10.1097/MPG.0000000000003716. Epub 2023 Feb 2. PMID 36735394